CLINICAL TRIAL: NCT07366957
Title: Determination of Motor Competence and Physical Activity Levels in Children Aged 4-6 and Their Relationship With Parental Perceptions: A Qualitative Study
Brief Title: Motor Competence and Physical Activity in Children Aged 4-6: Associations With Parental Perceptions
Status: Active, not recruiting | Type: Observational
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Server ERDOĞMUŞ, Msc. PT. / Research Assistant, Mudanya University
Other Study IDs: 2025/15-804
Record Dates: First submitted 2026-01-16; First posted 2026-01-26 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Motor Development; Physical Activity
Keywords: Motor competence; Motor development; Physical activity; Preschool children; Parental perceptions; Qualitative research
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 4-6 Years Old Children and Their Parents: This cohort includes typically developing children aged 4-6 years and their parents. Children's motor skills will be assessed using the Peabody Developmental Motor Scales - II (PDMS-II), and parents' perceptions of their children's motor abilities and physical activity will be evaluated through semi-structured interviews. No interventions or treatments will be applied.

SUMMARY:
This study aims to determine motor competence and physical activity levels in children aged 4-6 years and to explore their relationship with parental perceptions. The study will use a qualitative research approach supported by quantitative assessments. Children's motor competence will be evaluated using the Peabody Developmental Motor Scales-Second Edition (PDMS-II), while parents will participate in semi-structured interviews to explore their perceptions, attitudes, and experiences related to their children's motor development and physical activity. Data will be collected in educational settings without any intervention. The findings are expected to contribute to a better understanding of family-related factors influencing motor development in early childhood.

DETAILED DESCRIPTION:
This observational study aims to examine motor competence and physical activity levels in children aged 4-6 years and to explore their relationship with parental perceptions. Early childhood is a critical period for motor development, during which family-related factors may influence children's physical activity participation and motor skill acquisition.

The study will be conducted using a qualitative-dominant mixed-methods design with an embedded quantitative component. Children's motor competence will be assessed using the Peabody Developmental Motor Scales-Second Edition (PDMS-II), a standardized and validated tool for evaluating gross and fine motor skills in young children. Quantitative motor assessment data will be used to support and contextualize qualitative findings.

Parental perceptions will be explored through semi-structured interviews conducted separately with mothers and fathers. Interviews will focus on parents' views regarding their children's motor abilities, physical activity participation, and factors influencing these behaviors. Interviews will be conducted face-to-face, audio-recorded with participant consent, and transcribed verbatim for analysis.

The study will be carried out in educational settings in Bursa and Afyonkarahisar provinces. Participation will be voluntary, and written informed consent will be obtained from all parents prior to data collection. No interventions or experimental procedures will be applied during the study.

Quantitative data will be analyzed descriptively, while qualitative data will be analyzed using thematic analysis to identify key themes related to parental perceptions. Integration of quantitative and qualitative findings is expected to provide a comprehensive understanding of the relationship between motor competence, physical activity, and family perceptions in early childhood. The results may inform family-centered approaches in child health, education, and rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

Children

* Children aged 4-6 years based on chronological age,
* Children without any physician-diagnosed physical, intellectual, or neurological disorders,
* Children born at term (≥37 weeks of gestation),
* Children with no history of serious perinatal or postnatal complications (e.g., prolonged neonatal intensive care unit stay, intracranial hemorrhage, requirement for advanced respiratory support),
* Children able to independently complete the motor assessment tests used in the study.

Parents

* Parents who voluntarily agree to participate in the study and provide written informed consent,
* Parents with sufficient proficiency in reading, understanding, and expressing -themselves in Turkish,
* Parents who are the primary caregivers of the child included in the study.

Exclusion Criteria:

Children

* Children younger than 4 years or older than 6 years,
* Children with a history of preterm birth (<37 weeks of gestation),
* Children with any physician-diagnosed neurological, physical, developmental, or chronic conditions (e.g., cerebral palsy, pervasive developmental disorders, genetic syndromes, musculoskeletal disorders),
* Children with congenital or acquired orthopedic conditions that prevent completion of the motor tests used in the study,
* Children with attention, behavioral, or communication difficulties that would prevent completion of the test procedures.

Parents

* Individuals who have difficulty communicating in Turkish or are unable to participate in the interview process,
* Parents who do not complete the interview process, do not consent to audio recording, or voluntarily withdraw from the study were defined as exclusion criteria.

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: This study population consists of children aged 4-6 years who were born at term (≥37 weeks of gestation) and do not have any physician-diagnosed neurological, physical, or developmental conditions, along with their parents who serve as the primary caregivers. The study includes children who are able to independently perform the motor assessment tests and parents who voluntarily agree to participate, provide written informed consent, and are able to communicate in Turkish.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2026-01-10 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-03 (Estimated)

PRIMARY OUTCOMES:
Motor Development Scores (PDMS-II) | 12/2025-04/2026
  Children's gross and fine motor skills will be assessed using the Peabody Developmental Motor Scales - Second Edition (PDMS-II). The PDMS-II consists of gross motor and fine motor subtests and yields standard scores and composite scores.
  Raw scores are converted to standard scores, with a possible score range of 1 to 20 for subtests, and composite motor quotients ranging from 35 to 165.
  Higher scores indicate better motor performance and more advanced motor development.
  This measure provides objective and standardized data on motor development in children aged 4-6 years.

SECONDARY OUTCOMES:
Parental Perception Scores | 12/2025-04/2026
  Parents' perceptions and attitudes regarding their children's motor skills and participation in physical activity will be explored using semi-structured interviews.
  This outcome measure is qualitative in nature and does not involve a standardized scale or numerical scoring system.
  Interview data will be analyzed using thematic qualitative analysis to identify key themes related to parental understanding, perceptions, and support.
Parent-Child Motor Skill Concordance | 12/2025-04/2026
  The relationship between parental perceptions and children's actual PDMS-II motor scores will be examined using correlation analyses to explore discrepancies or alignments.

CONTACTS AND LOCATIONS:
Locations (1):
- Mudanya University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation/Afyonkarahisar University of Health Sciences - Atatürk Vocational School of Health Services - Physiotherapy Program, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No